CLINICAL TRIAL: NCT01921257
Title: A Multi-Centre, Single-Blind Study to Assess the Safety of Cat-PAD in Cat Allergic Paediatric Subjects
Brief Title: Paediatric Safety Study in Cat-PAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Collaborators: inVentiv Health Clinical (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CP009
Record Dates: First submitted 2013-07-17; First posted 2013-08-13 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Rhinoconjunctivitis
Keywords: Cat Allergy; Rhinoconjunctivitis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Cat-PAD and Placebo
  Interventions: Drug: Cat-PAD; Drug: Placebo

INTERVENTIONS:
Drug: Cat-PAD
Drug: Placebo

SUMMARY:
Study to Assess the Safety of Cat-PAD in Cat Allergic Paediatric Subjects

ELIGIBILITY:
* Inclusion Criteria

  * Male or female, aged 5-12 years.
  * Moderate to severe rhinoconjunctivitis on exposure to cats for at least 2 years.
  * Subjects may optionally also have GINA Step 1 controlled asthma.
  * Positive skin prick test to cat hair.
  * Cat dander specific IgE ≥0.35 kU/L.
* Exclusion Criteria

  * Asthma falling under the GINA definitions "partly controlled" and "uncontrolled" or Steps 2 to 5.
  * FEV1 <80% of predicted.
  * Clinically relevant abnormalities detected on physical examination.
  * History of severe drug allergy, severe angioedema or anaphylactic reaction to food.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Poland (3):
  - Lodz
  - Tarnów
  - Warsaw

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo run-in Followed by Cat-PAD: All participants; received two intradermal doses of placebo (saline) followed by eight intradermal administrations of Cat-PAD.
Period: Overall Study
Arm/Group | Placebo run-in Followed by Cat-PAD
Started | 16
Placebo run-in | 16
Active Treatment | 13
Completed | 13
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Study Participants: Overall study participants
Arm/Group | Study Participants
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Poland | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With AEs
Description: To evaluate the safety and tolerability of Cat-PAD in paediatric subjects aged 5 to <12 years.
Time Frame: up to 36 weeks after start of treatment
Population: All subjects enrolled
Measure: Number; unit: participants
Arm/Group | Study Participants
Number analyzed (Participants) | 16
participants
  Adverse Events Placebo | 5
  Adverse Events Cat-PAD | 12

ADVERSE EVENTS:
Time Frame: Overall study (up to 36 weeks after the start of treatment)
Groups:
- Placebo run-in: Placebo run-in
- Cat-PAD: Active treatment (Cat-PAD)
Arm/Group | Placebo run-in | Cat-PAD
Serious Adverse Events (participants affected / at risk) | 0/16 | 2/16
Other Adverse Events (participants affected / at risk) | 5/16 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo run-in (N=16) | Cat-PAD (N=16)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo run-in (N=16) | Cat-PAD (N=16)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Allergy to animal (Immune system disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (7)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 5 (8)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Laryngitis (Infections and infestations) | 0 (0) | 2 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
To avoid disclosures that may affect the proprietary rights of the Sponsor, the Investigator agrees to allow Circassia the opportunity to review all manuscripts and abstracts 60 days prior to submission for publication. Circassia reserves the right to include the report of this study in any regulatory documentation or submission or in any informational materials.